CLINICAL TRIAL: NCT02554084
Title: Optical Coherence Tomography of Tear Film Dynamics In-Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jannick Rolland-Thompson, Professor, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 52165
Record Dates: First submitted 2014-11-24; First posted 2015-09-18 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Eye Disease (Experimental): Optical Coherence Tomography
  Interventions: Other: Optical Coherence Tomography
- Normals (Active Comparator): Optical Coherence Tomography
  Interventions: Other: Optical Coherence Tomography

INTERVENTIONS:
Other: Optical Coherence Tomography — Digital images of tear film

SUMMARY:
The purpose of this study is to evaluate a new instrument that takes digital images of tear film (a thin film that coats the eye that is made up of oil and water). The investigators are interested in measuring how the thickness of the tear film varies through time. The goal is to develop a technique that may enable non-invasive evaluation of Dry Eye Disease for future clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed Dry Eye Disease
* Normal individuals (those without a dry eye diagnosis and without eye abnormalities)
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study
* Either gender
* Any racial or ethnic origin

Exclusion Criteria:

* Use of any prescription ocular medication (such as but not limited to, glaucoma medications and Restasis) used within 14 days of the study visit
* Current eye disease, infection or inflammation that affects the surface of the eye such as, but not limited to blepharitis and ocular allergy
* Past eye surgery, such as, but not limited to, refractive surgery. Subjects who have had cataract surgery less than one year ago
* Use of soft or hard contact lenses 6 hours prior to visit
* Female subjects may not be pregnant or lactating (subjects will be asked to self-report these conditions)
* Infectious diseases (for example, hepatitis, tuberculosis) or an immuno-suppressive disease (for example, HIV) (subjects will be asked to self-report these conditions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Thickness of lipid layers on patient cornea (nm) | participants will be seen once within a one year period, on average within 1 month
  Multiple measures taken within one eye blink, through optical coherence tomography, to map thickness. Each individual measure taken contributes to a computed map of lipid-layer thickness.
Thickness of aqueous layers on patient cornea (um) | participants will be seen once within a one year period, on average within 1 month
  Multiple measures taken within one eye blink, through optical coherence tomography, to map thickness. Each individual measure taken contributes to a computed map of aqueous-layer thickness.

SECONDARY OUTCOMES:
Thickness maps dynamics | participants will be seen once within a one year period, on average within 1 month
  Measured through optical coherence tomography
Optical aberrations | participants will be seen once within a one year period, on average within 1 month
  Measured through optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Jannick Rolland, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States